CLINICAL TRIAL: NCT03846713
Title: Effect of Thermal-softening of Double-lumen Endobronchial Tubes on Success Rate of Airway Exchange Catheter
Brief Title: Thermosoftening of Double-lumen Tube for Airway Exchanger Catheter
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jae-Hyon Bahk, MD, PhD, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: JHBahk_DLT_AEC
Record Dates: First submitted 2019-01-09; First posted 2019-02-20 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Intubation Complication; Hoarseness; Sore Throat
Keywords: double-lumen tube; intubation; airway exchange catheter; thermosoftening
MeSH Terms: conditions — Hoarseness; Pharyngitis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- non-thermosoftening (Active Comparator): Double-lumen tube is put into a bottle of normal saline at room temperature (25°C) before intubation.
  Interventions: Procedure: non-thermosoftening
- thermosoftening (Experimental): Double-lumen tube is put into a bottle of warm normal saline (40°C) before intubation.
  Interventions: Procedure: thermosoftening

INTERVENTIONS:
Procedure: non-thermosoftening — By using airway exchange catheter, tube exchange is performed from single to double lumen tube that was put into normal saline at room temperature.
  Arms: non-thermosoftening
Procedure: thermosoftening — By using airway exchange catheter, tube exchange is performed from single to double lumen tube that was put into warm normal saline (40°C).
  Arms: thermosoftening

SUMMARY:
The purpose of this study is to investigate the effect of double-lumen tube thermal-softening before intubation on the success rate of tube exchange by airway exchange catheter.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing thoracic surgery that requires bronchoscopy study before the placement of double-lumen tubes

Exclusion Criteria:

* Preoperative hoarseness or a sore throat
* History of upper airway diseases
* Anticipated difficult airway

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2017-12-27 (Actual); Primary Completion 2019-03-31 (Actual); Study Completion 2019-05-31 (Actual)

PRIMARY OUTCOMES:
Time to intubate | Intraoperative (During exchanging single- to double-lumen tube)
  Length of time to exchange endotracheal tube from single- to double-lumen tube using airway exchange catheter.

SECONDARY OUTCOMES:
Postoperative hoarseness (4-points scoring) | up to 48 hours after surgery
postoperative sore throat (4-points scoring) | up to 48 hours after surgery
Vocal cord injuries assessed by videolaryngoscope | up to 1 hour after double-lumen tube extubation
  vocal cord injuries observed after tube-exchange

CONTACTS AND LOCATIONS:
Overall Officials: Jae-Hyon Bahk, MD, PhD, Study Chair — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, Seoul, South Korea